CLINICAL TRIAL: NCT04013425
Title: Socket Preservation Using the Ice Cream Cone Technique Versus Spontaneous Healing in Fresh Extraction Sockets.
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Andrew George Edward Aziz, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Philo new protocol
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Socket Preservation
Keywords: Socket preservation; Alveolar Ridge Preservation; Ridge Preservation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice Cream Cone Technique (Experimental): Atraumatic extraction followed by addition of barrier membrane and xenograft in the socket.
  Interventions: Procedure: Ice Cream Cone Technique
- Spontaneous Healing (No Intervention): Spontaneous Healing after Atraumatic Extraction

INTERVENTIONS:
Procedure: Ice Cream Cone Technique — Guided bone regeneration
  Arms: Ice Cream Cone Technique

SUMMARY:
The research is about socket preservation using the ice cream cone technique including collagen membrane and xenograft compared to spontaneous healing.

DETAILED DESCRIPTION:
Atraumatic extraction is done and the socket is either left for spontaneous healing or the ice cream cone technique using the collagen membrane and the socket is filled with xenograft.

ELIGIBILITY:
Inclusion Criteria:

* Single or double rooted teeth indicated for extraction
* Presence of a buccal defect.
* Maxillary and Mandibular Arches

Exclusion Criteria:

* Systemic conditions/disease that contraindicated surgery.
* Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.
* Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.
* Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Horizontal Bone Dimension from the CBCT in mm. | 3 months
  from the CBCT in mm.

SECONDARY OUTCOMES:
Buccal Vertical Bone Dimension | 3 months
  from CBCT in mm.
Palatal Vertical Bone Dimension | 3 months
  from CBCT in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrew George, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tan-Chu JH, Tuminelli FJ, Kurtz KS, Tarnow DP. Analysis of buccolingual dimensional changes of the extraction socket using the "ice cream cone" flapless grafting technique. Int J Periodontics Restorative Dent. 2014 May-Jun;34(3):399-403. doi: 10.11607/prd.1605. PMID 24804291